CLINICAL TRIAL: NCT02559622
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Exploratory Evaluation of Surrogate Markers of Cardiovascular Risk in Patients With Active Chronic Plaque-type Psoriasis Treated for up to 52 Weeks With Subcutaneous (s.c.) Secukinumab (300 mg or 150 mg).
Brief Title: Evaluation of Cardiovascular Risk Markers in Psoriasis Patients Treated With Secukinumab
Acronym: CARIMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457ADE02
Record Dates: First submitted 2015-08-04; First posted 2015-09-24 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 300 mg secukinumab (Experimental): 300 mg secukinumab every week for 4 weeks followed by 300 mg secukinumab every 4 weeks until week 48 (last injection)
  Interventions: Drug: Secukinumab
- 150 mg secukinumab (Experimental): 150 mg secukinumab every week for 4 weeks followed by 150 mg secukinumab every 4 weeks until week 48 (last injection)
  Interventions: Drug: Secukinumab
- Placebo followed by 300 mg secukinumab (Other): Placebo until week 12 followed by 300 mg secukinumab every week for 4 weeks followed by 300 mg secukinumab every 4 weeks until week 48 (last injection)
  Interventions: Other: Placebo
- Placebo followed by 150 mg secukinumab (Other): Placebo until week 12 followed by 150 mg secukinumab every week for 4 weeks followed by 150 mg secukinumab every 4 weeks until week 48 (last injection)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Secukinumab — 300 mg secukinumab
  Other Names: AIN457
  Arms: 300 mg secukinumab
Other: Placebo — Placebo followed by 300 mg secukinumab
  Arms: Placebo followed by 300 mg secukinumab
Other: Placebo — Placebo followed by 150 mg secukinumab
  Arms: Placebo followed by 150 mg secukinumab
Drug: Secukinumab — 150 mg secukinumab
  Other Names: AIN457
  Arms: 150 mg secukinumab

SUMMARY:
The purpose of this study was to explore the effect of treatment with 300 mg or with 150 mg secukinumab (administered weekly for 4 weeks followed by four-weekly administration) on endothelial dysfunction and arterial stiffness after 12 weeks and for up to 52 weeks in subjects with chronic plaque-type psoriasis. Furthermore soluble biomarkers were assessed to evaluate the influence of secukinumab on cardiovascular risk. Magnetic resonance imaging (MRI) was performed in a sub-population to assess the treatment effect on arterial vessel wall morphometry in atherosclerosis prone vascular beds.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic moderate to severe plaque type psoriasis for at least 6 months prior to randomization with a Psoriasis Area and Severity Index (PASI) score ≥ 10 at randomization.
* Inadequate response, intolerance or contraindication to cyclosporine, methotrexate and psoralen plus ultraviolet A light treatment (PUVA) as documented in the patient's medical history or reported by the patient or determined by the investigator at screening. Relative contraindications such as interference of patient's lifestyle with the treatment are accepted.

Key Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and guttata psoriasis) at screening or randomization.
* Ongoing use of prohibited psoriasis and non-psoriasis treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- Germany (22):
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Langenau
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Ulm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 23 centers in Germany.
Groups:
- Secukinumab 300 mg: Participants were administered with 300 milligrams (mg) secukinumab subcutaneously (s.c.) using pre-filled syringe every week for 4 weeks followed by 300 mg secukinumab every 4 weeks until week 48 (last injection).
- Secukinumab 150 mg: Participants were administered with 150 mg secukinumab s.c. using pre-filled syringe every week for 4 weeks followed by 150 mg secukinumab every 4 weeks until week 48 (last injection).
- Placebo Followed by 300 mg Secukinumab: Participants were administered with placebo until week 12 followed by 300 mg secukinumab s.c. using pre-filled syringe every week for 4 weeks followed by 300 mg secukinumab every 4 weeks until week 48 (last injection).
- Placebo Followed by 150 mg Secukinumab: Participants were administered with placebo until week 12 followed by 150 mg secukinumab s.c. using pre-filled syringe every week for 4 weeks followed by 150 mg secukinumab every 4 weeks until week 48 (last injection).
Period: Overall Study
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Started | 48 | 54 | 26 | 23
Completed | 47 | 49 | 24 | 20
Not Completed | 1 | 5 | 2 | 3
Not completed — Progressive disease | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 2 | 2
Not completed — Patient/guardian decision | 1 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Secukinumab 300 mg: Participants were administered with 300 mg secukinumab s.c. using pre-filled syringe every week for 4 weeks followed by 300 mg secukinumab every 4 weeks until week 48 (last injection).
- Total: Total of all reporting groups
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab | Total
Number analyzed (Participants) | 48 | 54 | 26 | 23 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 46 | 46 | 26 | 22 | 140
  >=65 years | 2 | 8 | 0 | 1 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (12.9) | 46.0 (14.4) | 43.7 (11.4) | 46.8 (13.1) | 45.2 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 23 | 8 | 7 | 49
  Male | 37 | 31 | 18 | 16 | 102
Region of Enrollment [Number; unit: participants]
  Germany | 48 | 54 | 26 | 23 | 151

OUTCOME MEASURES:

1. Primary Outcome: Flow Mediated Dilation (FMD) at Week 12 Followed by Secukinumab 300 mg vs Pooled Placebo Treatment
Description: Flow Mediated Dilation (FMD) is non-invasive method evaluated by Doppler Ultrasound test, to assess endothelial function. FMD was calculated as the percent maximal deviation from the baseline arterial diameter (D):FMD = 100*[(D maximum - D baseline) / D baseline]. Here, arterial diameter (brachial artery) was measured at rest (1 minute), during inflation of the distal cuff to 100 millimeter of mercury (mmHg) for 4.5 minutes and for 4.5 minutes following deflation.
Time Frame: Week 12
Population: The analysis was performed in Full analysis set (FAS) population, defined as all participants from the randomized set who received at least one dose of study drug. Here, "Number analyzed" signifies participants evaluable for FMD at Week 12 for each arm, respectively.
Measure: Mean (Standard Deviation); unit: Percentage maximal increase in diameter
Groups:
- Placebo (Pooled): Participants were administered with placebo until week 12 followed by 150 mg or 300 mg secukinumab s.c. using pre-filled syringe every week for 4 weeks followed by 150 mg or 300 mg secukinumab respectively every 4 weeks until week 48 (last injection).
Arm/Group | Secukinumab 300 mg | Placebo (Pooled)
Number analyzed (Participants) | 39 | 38
Percentage maximal increase in diameter | 5.23 (5.30) | 3.65 (4.07)
Statistical Analysis 1: Comparison: Secukinumab 300 mg vs Placebo (Pooled); Test type: Superiority; p = 0.2230, ANCOVA; Least Square (LS) mean difference = 1.17, 95% CI 2-sided [-0.72 to 3.06]

2. Secondary Outcome: Change From Baseline in Flow Mediated Dilation (FMD) at Week 4, 12, 24 and 52
Description: FMD is non-invasive method evaluated by Doppler Ultrasound test, to assess endothelial function. FMD was calculated as the percent maximal deviation from the baseline arterial diameter (D):FMD = 100*[(D maximum - D baseline) / D baseline]. Here, arterial diameter (brachial artery) was measured at rest (1 minute), during inflation of the distal cuff to 100 mmHg for 4.5 minutes and for 4.5 minutes following deflation. A positive change in FMD constitutes an improvement in endothelial function.
Time Frame: Baseline, Week 4, 12, 24 and 52
Population: The analysis was performed in FAS population. Here, "Number analyzed" signifies participants evaluable for FMD at weeks 4, 12, 24 and 52 for each arm, respectively.
Measure: Mean (95% Confidence Interval); unit: Percentage change in FMD
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Number analyzed (Participants) | 48 | 54 | 26 | 23
Percentage change in FMD
  Week 4: number analyzed (Participants) | 37 | 47 | 21 | 16
  Week 4 | -0.7 [-1.9 to 0.5] | -0.9 [-2.4 to 0.7] | 0.7 [-1.0 to 2.5] | 1.4 [-0.8 to 3.6]
  Week 12: number analyzed (Participants) | 39 | 48 | 21 | 17
  Week 12 | 0.5 [-1.1 to 2.1] | 0.1 [-1.2 to 1.5] | -0.1 [-2.7 to 2.4] | 0.1 [-2.1 to 2.3]
  Week 24: number analyzed (Participants) | 35 | 39 | 19 | 16
  Week 24 | -0.8 [-1.9 to 0.3] | 1.0 [-0.4 to 2.4] | -0.0 [-2.6 to 2.6] | 0.9 [-1.0 to 2.9]
  Week 52: number analyzed (Participants) | 38 | 43 | 20 | 17
  Week 52 | 2.1 [0.8 to 3.3] | 2.1 [0.7 to 3.4] | 2.2 [-0.5 to 4.9] | 1.2 [-1.0 to 3.5]

3. Secondary Outcome: Change From Baseline in Aortic Augmentation Index at Heart Rate of 75 (AIx-75) at Week 4, 12, 24 and 52
Description: Pulse wave analysis was performed on the central aortic pressure waveform as derived by SphygmoCor XCEL from the brachial pressure waveform recorded in a partially-inflated blood pressure cuff around the upper arm. The waveform derivation employs a validated generalized transfer function to convert a brachial waveform to a central waveform and has been shown to produce measurement results corresponding to measurements using intra-arterial pressure catheters. The augmentation index is derived from the waveform by determining the percentage of the central pulse pressure during systole due to wave reflection. AIx was heart-rate corrected to calculate the AIx at a heart rate of 75 bpm, i.e. AIx-75.
Time Frame: Baseline, Week 4, 12, 24 and 52
Population: The analysis was performed in FAS population. Here, "Number analyzed" signifies participants evaluable for pulse wave analysis at weeks 4, 12, 24 and 52 for each arm, respectively.
Measure: Mean (95% Confidence Interval); unit: Percentage change in Alx-75
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Number analyzed (Participants) | 48 | 54 | 26 | 23
Percentage change in Alx-75
  Week 4: number analyzed (Participants) | 47 | 52 | 25 | 21
  Week 4 | 0.0 [-2.8 to 2.9] | 0.3 [-2.0 to 2.7] | 1.1 [-1.7 to 3.8] | -0.1 [-3.0 to 2.9]
  Week 12: number analyzed (Participants) | 48 | 52 | 26 | 21
  Week 12 | -0.5 [-3.0 to 2.1] | 1.0 [-1.7 to 3.8] | -1.1 [-5.4 to 3.3] | -0.1 [-3.4 to 3.2]
  Week 24: number analyzed (Participants) | 47 | 50 | 24 | 21
  Week 24 | 3.0 [0.3 to 5.6] | 1.8 [-0.6 to 4.3] | 1.3 [-2.7 to 5.3] | 0.7 [-2.7 to 4.1]
  Week 52: number analyzed (Participants) | 47 | 49 | 25 | 20
  Week 52 | 1.3 [-1.5 to 4.2] | -0.1 [-2.8 to 2.7] | -1.4 [-5.8 to 2.9] | -0.9 [-4.2 to 2.5]

4. Secondary Outcome: Change From Baseline in Pulse Wave Velocity (PWV) at Week 4, 12, 24 and 52
Description: Regional arterial pulse wave velocity (PWV) was directly related to arterial stiffness and was defined as the time it takes for the blood pressure wave to travel from a proximal site to a distal site (relative to the heart) divided by the distance (PWV = ∆distance/∆time [m/s]). The foot of the arterial pulse wave was being recorded by using the SphygmoCor XCEL device. XCEL simultaneously measures the pressure waveform at the femoral site (using a partially inflated custom blood pressure cuff) and the carotid site (using hand-held applanation tonometry). The foot-to-foot time between the two pressure waveforms was the time interval used in the PWV calculation.
Time Frame: Baseline, Week 4, 12, 24 and 52
Population: The analysis was performed in FAS population. Here, "n" signifies the sum of participants for all repeated measurements during calculation of mean, evaluable for pulse wave velocity (PWV) at Week 4, 12, 24 and 52 for each arm, respectively.
Measure: Mean (95% Confidence Interval); unit: meters per second (m/s)
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Number analyzed (Participants) | 48 | 54 | 26 | 23
meters per second (m/s)
  Week 4 (n = 192, 262, 133, 104) | 0.0 [-0.2 to 0.2] | -0.2 [-0.3 to 0.0] | 0 [-0.1 to 0.2] | -0.2 [-0.5 to 0.2]
  Week 12 (n = 214, 255, 116, 133) | 0.4 [0.2 to 0.6] | 0.1 [-0.1 to 0.2] | 0.1 [-0.2 to 0.4] | 0.4 [0.1 to 0.7]
  Week 24 (n = 205, 255, 100, 100) | 0.2 [-0.1 to 0.5] | 0.0 [-0.2 to 0.1] | 0.2 [0.1 to 0.4] | -0.1 [-0.5 to 0.2]
  Week 52 (n = 191, 228, 115, 101) | -0.1 [-0.3 to 0.0] | 0.2 [-0.1 to 0.5] | 0.1 [-0.2 to 0.4] | -0.2 [-0.6 to 0.2]

5. Secondary Outcome: Change From Baseline in Average Wall Area Assessed as a Measure of Total Plaque Burden at Week 12
Description: Magnetic resonance imaging (MRI) was used to evaluate vessel wall morphometry to determine plaque burden. As a measure of plaque burden, average wall area was computed by subtracting vessel lumen area from total vessel area. Exploratory 3.0 Tesla MRI technique was applied to assess structure and function of the carotid and the aorta. A 2D axial dark blood T1, T2, proton density weighted spin echo based images and time of flight images were acquired from the bilateral carotid arteries as well as the descending aorta.
Time Frame: Baseline, Week 12
Population: The analysis was performed in FAS population. Here, "Number analyzed" signifies participants evaluable for MRI sub-study at week 12 for each arm, respectively. MRI was applied in a sub-study population of 33 participants.
Measure: Mean (95% Confidence Interval); unit: millimeter square (mm^2)
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Number analyzed (Participants) | 48 | 54 | 26 | 23
millimeter square (mm^2)
  Ascending thoracic aorta: number analyzed (Participants) | 10 | 11 | 4 | 6
  Ascending thoracic aorta | 15.35 [-8.23 to 38.92] | 5.91 [-13.09 to 24.91] | 9.92 [-58.24 to 78.08] | 6.45 [-9.26 to 22.15]
  Descending thoracic aorta: number analyzed (Participants) | 10 | 11 | 4 | 7
  Descending thoracic aorta | 2.69 [-14.18 to 19.56] | -2.94 [-13.44 to 7.57] | -4.04 [-29.61 to 21.53] | 3.16 [-13.73 to 20.05]
  Carotid bifurcation left: number analyzed (Participants) | 11 | 11 | 4 | 7
  Carotid bifurcation left | 0.52 [-2.72 to 3.77] | -1.08 [-3.85 to 1.69] | 3.63 [-7.82 to 15.08] | 1.12 [-2.04 to 4.28]
  Carotid bifurcation right: number analyzed (Participants) | 11 | 11 | 4 | 7
  Carotid bifurcation right | -0.77 [-3.60 to 2.06] | 1.75 [-0.71 to 4.21] | -1.26 [-7.64 to 5.12] | -1.07 [-4.24 to 2.10]
  Common carotid left: number analyzed (Participants) | 11 | 11 | 4 | 6
  Common carotid left | 0.17 [-1.64 to 1.99] | 1.12 [-1.80 to 4.03] | 0.69 [-5.21 to 6.59] | 0.12 [-1.91 to 2.15]
  Common carotid right: number analyzed (Participants) | 11 | 11 | 4 | 7
  Common carotid right | -0.12 [-2.17 to 1.92] | 0.30 [-2.76 to 3.36] | -0.38 [-6.56 to 5.80] | -0.14 [-1.60 to 1.32]
  Internal carotid left: number analyzed (Participants) | 9 | 10 | 4 | 5
  Internal carotid left | 3.79 [-0.19 to 7.78] | 2.09 [-0.57 to 4.75] | 2.59 [-0.58 to 5.77] | -1.74 [-4.55 to 1.08]
  Internal carotid right: number analyzed (Participants) | 11 | 11 | 4 | 7
  Internal carotid right | -0.69 [-1.90 to 0.51] | 0.17 [-1.96 to 2.30] | 0.68 [-3.97 to 5.33] | -1.37 [-4.37 to 1.62]
  Descending abdominal aorta: number analyzed (Participants) | 8 | 9 | 4 | 6
  Descending abdominal aorta | 8.71 [-6.33 to 23.76] | -3.79 [-21.90 to 14.32] | 4.56 [-52.64 to 61.77] | -0.58 [-15.51 to 14.35]

6. Secondary Outcome: Change From Baseline in Average Wall Area Assessed as a Measure of Total Plaque Burden at Week 52
Description: as for outcome 5
Time Frame: Baseline, Week 52
Population: The analysis was performed in FAS population. Here, "Number analyzed" signifies participants evaluable for MRI sub-study at week 52 for each arm, respectively. MRI was applied in a sub-study population of 33 participants.
Measure: Mean (95% Confidence Interval); unit: mm^2
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Number analyzed (Participants) | 48 | 54 | 26 | 23
mm^2
  Ascending thoracic aorta: number analyzed (Participants) | 10 | 11 | 4 | 6
  Ascending thoracic aorta | 14.42 [-14.93 to 43.76] | 3.19 [-17.17 to 23.55] | -15.11 [-28.15 to -2.06] | 9.54 [-14.71 to 33.79]
  Descending thoracic aorta: number analyzed (Participants) | 10 | 11 | 4 | 7
  Descending thoracic aorta | 3.97 [-13.42 to 21.37] | 2.55 [-12.23 to 17.33] | -10.14 [-34.05 to 13.77] | 1.14 [-26.76 to 29.05]
  Carotid bifurcation left: number analyzed (Participants) | 11 | 11 | 4 | 7
  Carotid bifurcation left | 2.45 [-1.55 to 6.45] | 0.64 [-3.59 to 4.88] | 0.58 [-9.03 to 10.20] | 2.60 [-2.16 to 7.36]
  Carotid bifurcation right: number analyzed (Participants) | 11 | 11 | 4 | 7
  Carotid bifurcation right | -1.64 [-6.02 to 2.74] | -0.05 [-3.62 to 3.51] | -3.23 [-9.86 to 3.40] | 1.25 [-3.92 to 6.41]
  Common carotid left: number analyzed (Participants) | 11 | 11 | 4 | 6
  Common carotid left | 1.42 [-0.36 to 3.19] | 1.21 [-1.51 to 3.93] | 0.65 [-2.82 to 4.13] | 1.00 [-0.83 to 2.82]
  Common carotid right: number analyzed (Participants) | 11 | 11 | 4 | 7
  Common carotid right | 0.02 [-2.54 to 2.58] | 0.23 [-2.29 to 2.75] | -0.80 [-6.25 to 4.64] | -1.38 [-3.33 to 0.57]
  Internal carotid left: number analyzed (Participants) | 9 | 10 | 4 | 5
  Internal carotid left | 5.43 [1.21 to 9.65] | 3.59 [0.59 to 6.60] | 1.06 [-2.66 to 4.78] | 0.33 [-5.07 to 5.73]
  Internal carotid right: number analyzed (Participants) | 11 | 11 | 4 | 7
  Internal carotid right | -1.07 [-2.12 to -0.03] | 0.71 [-1.78 to 3.21] | -0.20 [-3.89 to 3.49] | 0.13 [-2.22 to 2.48]
  Descending abdominal aorta: number analyzed (Participants) | 8 | 9 | 4 | 6
  Descending abdominal aorta | 10.56 [-8.37 to 29.48] | -4.36 [-17.90 to 9.19] | 12.46 [-46.12 to 71.05] | 11.82 [-15.26 to 38.90]

7. Secondary Outcome: Change From Baseline in High Sensitivity C-reactive Protein (hsCRP) at Week 4, 12, 24 and 52
Description: High sensitivity C-reactive protein (hsCRP), a soluble biomarker of systemic inflammation was determined in fasting blood samples to evaluate the effect of secukinumab on systemic inflammation.
Time Frame: Baseline, Week 4, 12, 24 and 52
Population: The analysis was performed in FAS population. Here, "Number analyzed" signifies participants evaluable for hsCRP at week 4, 12, 24 and 52 for each arm, respectively.
Measure: Mean (95% Confidence Interval); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Number analyzed (Participants) | 48 | 54 | 26 | 23
Milligrams per deciliter (mg/dL)
  Week 4: number analyzed (Participants) | 48 | 53 | 26 | 21
  Week 4 | 0.0 [-0.2 to 0.2] | -0.2 [-0.4 to -0.1] | -0.0 [-0.2 to 0.2] | 0.1 [-0.1 to 0.3]
  Week 12: number analyzed (Participants) | 48 | 54 | 26 | 21
  Week 12 | -0.0 [-0.3 to 0.3] | -0.2 [-0.3 to 0.0] | -0.3 [-0.8 to 0.1] | 0.1 [-0.4 to 0.6]
  Week 24: number analyzed (Participants) | 48 | 52 | 25 | 21
  Week 24 | -0.0 [-0.3 to 0.2] | -0.0 [-0.3 to 0.2] | 0.1 [-0.2 to 0.4] | -0.4 [-0.9 to 0.1]
  Week 52: number analyzed (Participants) | 48 | 50 | 26 | 20
  Week 52 | -0.1 [-0.3 to 0.1] | -0.2 [-0.4 to -0.0] | -0.3 [-0.8 to 0.2] | -0.5 [-1.1 to 0.0]

8. Secondary Outcome: Change From Baseline in S-100 Protein B (Total) at Week 4, 12, 24 and 52
Description: S100 calcium-binding protein B (S100B-protein), a soluble biomarker of systemic inflammation was determined in fasting blood samples to evaluate the effect of secukinumab on systemic inflammation.
Time Frame: Baseline, Week 4, 12, 24 and 52
Population: The analysis was performed in FAS population. Here, "Number analyzed" signifies participants evaluable for S100B-protein at week 4, 12, 24 and 52 for each arm, respectively.
Measure: Mean (95% Confidence Interval); unit: Microgram per Liter (ug/L)
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Number analyzed (Participants) | 48 | 54 | 26 | 23
Microgram per Liter (ug/L)
  Week 4: number analyzed (Participants) | 48 | 53 | 26 | 22
  Week 4 | -0.0 [-0.0 to -0.0] | -0.0 [-0.0 to 0.0] | 0.0 [-0.0 to 0.0] | 0.0 [-0.0 to 0.0]
  Week 12: number analyzed (Participants) | 48 | 52 | 26 | 22
  Week 12 | -0.0 [-0.0 to 0.0] | -0.0 [-0.0 to 0.0] | 0.0 [-0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Week 24: number analyzed (Participants) | 48 | 51 | 25 | 22
  Week 24 | -0.0 [-0.0 to 0.0] | 0.0 [-0.0 to 0.0] | 0.0 [-0.0 to 0.0] | 0.0 [-0.0 to 0.0]
  Week 52: number analyzed (Participants) | 48 | 51 | 26 | 22
  Week 52 | -0.0 [-0.0 to 0.0] | -0.0 [-0.0 to -0.0] | 0.0 [-0.0 to 0.0] | -0.0 [-0.0 to 0.0]

9. Secondary Outcome: Change From Baseline in Chemokine (C-c Motif) Ligand 5 (CCL5), Monocyte Chemoattractant Protein 1 (MCP-1) and Macrophage Inflammatory Proteins (MIP) 1 Alpha and 1 Beta at Week 4, 12, 24 and 52
Description: Chemokine (c-c motif) ligand 5 (CCL5), Monocyte chemoattractant protein 1 (MCP-1) and Macrophage inflammatory proteins (MIP) 1 alpha (1A) and 1 beta (1B), soluble biomarkers of systemic inflammation were determined in fasting blood samples to evaluate the effect of secukinumab on systemic inflammation.
Time Frame: Baseline, Week 4, 12, 24 and 52
Population: The analysis was performed in FAS population. Here, "Number analyzed" signifies participants evaluable for CCL5, MCP-1, MIP-1A and MIP-1B at week 4, 12, 24 and 52 for each arm, respectively.
Measure: Mean (95% Confidence Interval); unit: picograms per milliliter (pg/mL)
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Number analyzed (Participants) | 48 | 54 | 26 | 23
picograms per milliliter (pg/mL)
  CCL5 Week 4: number analyzed (Participants) | 48 | 54 | 26 | 22
  CCL5 Week 4 | -1000 [-3106 to 1094] | 1649 [-597 to 3895] | 27.0 [-3943 to 3997] | -2000 [-5056 to 281.3]
  CCL5 Week 12: number analyzed (Participants) | 48 | 54 | 26 | 22
  CCL5 Week 12 | 2116 [-2368 to 6599] | 5185 [840.3 to 9530] | 4393 [-1598 to 10383] | 3002 [-1806 to 7809]
  CCL5 Week 24: number analyzed (Participants) | 48 | 52 | 25 | 22
  CCL5 Week 24 | 7772 [3766 to 11777] | 10000 [6437 to 14394] | 11000 [2117 to 20176] | 9168 [2124 to 16212]
  CCL5 Week 52: number analyzed (Participants) | 48 | 51 | 25 | 22
  CCL5 Week 52 | 1515 [-2478 to 5507] | 3577 [-737 to 7891] | -597 [-3340 to 2145] | 2308 [-2558 to 7175]
  MCP-1 Week 4: number analyzed (Participants) | 48 | 54 | 26 | 22
  MCP-1 Week 4 | -7.0 [-21.8 to 7.7] | 1.4 [-17.4 to 20.2] | -25 [-57.2 to 8.0] | 17.5 [-43.1 to 78.0]
  MCP-1 Week 12: number analyzed (Participants) | 48 | 54 | 26 | 22
  MCP-1 Week 12 | 18.4 [-1.9 to 38.7] | 28.6 [-8.4 to 65.7] | 11.3 [-40.9 to 63.5] | 21.5 [-18.3 to 61.2]
  MCP-1 Week 24: number analyzed (Participants) | 48 | 52 | 25 | 22
  MCP-1 Week 24 | 39.8 [-0.6 to 80.3] | 241 [-203 to 685.7] | -20 [-53.9 to 14.2] | 33.4 [8.3 to 58.5]
  MCP-1 Week 52: number analyzed (Participants) | 48 | 51 | 25 | 22
  MCP-1 Week 52 | 22.1 [-18.1 to 62.4] | 25.4 [-21.7 to 72.6] | -11 [-60.6 to 38.6] | 109 [-13.3 to 230.9]
  MIP-1A Week 4: number analyzed (Participants) | 48 | 54 | 26 | 22
  MIP-1A Week 4 | -0.1 [-2.1 to 1.9] | 0.1 [-1.6 to 1.8] | 0.5 [-2.5 to 3.5] | -0.6 [-2.3 to 1.2]
  MIP-1A Week 12: number analyzed (Participants) | 48 | 54 | 26 | 22
  MIP-1A Week 12 | 0.2 [-2.8 to 3.3] | 2.2 [-1.0 to 5.3] | -3.6 [-7.0 to -0.3] | 0.9 [-3.0 to 4.8]
  MIP-1A Week 24: number analyzed (Participants) | 48 | 52 | 25 | 22
  MIP-1A Week 24 | -0.2 [-2.9 to 2.4] | -0.5 [-3.6 to 2.6] | -4.7 [-8.4 to -1.0] | 1.7 [-1.3 to 4.7]
  MIP-1A Week 52: number analyzed (Participants) | 48 | 51 | 25 | 22
  MIP-1A Week 52 | 4.3 [-0.1 to 8.7] | 0.8 [-3.0 to 4.5] | 1.7 [-6.0 to 9.5] | 20.1 [4.7 to 35.6]
  MIP-1B Week 4: number analyzed (Participants) | 48 | 54 | 26 | 22
  MIP-1B Week 4 | -24 [-50.8 to 3.0] | -2.6 [-24.8 to 19.5] | -16 [-57.5 to 25.8] | -20 [-54.4 to 15.3]
  MIP-1B Week 12: number analyzed (Participants) | 48 | 54 | 26 | 22
  MIP-1B Week 12 | -49 [-80.9 to -16.6] | -34 [-69.0 to 1.4] | -65 [-106 to -24.7] | -68 [-116 to -20.5]
  MIP-1B Week 24: number analyzed (Participants) | 48 | 52 | 25 | 22
  MIP-1B Week 24 | -52 [-130 to 26.7] | -97 [-133 to -61.3] | -161 [-207 to -114] | 79.4 [-261 to 420.3]
  MIP-1B Week 52: number analyzed (Participants) | 48 | 51 | 25 | 22
  MIP-1B Week 52 | -41 [-73.6 to -8.6] | -59 [-89.0 to -29.7] | -73 [-122 to -24.2] | -31 [-109 to 46.8]

10. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 4, 12, 24 and 52
Description: Fasting plasma glucose (FPG), a soluble biomarker of Dysglycemia was determined in fasting blood samples to evaluate the effect of secukinumab on systemic inflammation.
Time Frame: Baseline, Week 4, 12, 24 and 52
Population: The analysis was performed in FAS population. Here, "Number analyzed" signifies participants evaluable for FPG at week 4, 12, 24 and 52 for each arm, respectively.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Number analyzed (Participants) | 48 | 54 | 26 | 23
mg/dL
  Week 4: number analyzed (Participants) | 47 | 53 | 26 | 22
  Week 4 | 1.5 [-1.0 to 4.0] | -1.6 [-4.6 to 1.3] | 0.9 [-4.4 to 6.1] | 0.2 [-5.2 to 5.6]
  Week 12: number analyzed (Participants) | 47 | 53 | 26 | 22
  Week 12 | 3.5 [-0.0 to 7.0] | 1.1 [-4.0 to 6.2] | 5.3 [-2.2 to 12.8] | -1.5 [-7.1 to 4.0]
  Week 24: number analyzed (Participants) | 47 | 51 | 25 | 22
  Week 24 | 2.5 [0.0 to 5.0] | 1.4 [-6.3 to 9.1] | 12.1 [-10.8 to 35.0] | -1.4 [-7.7 to 5.0]
  Week 52: number analyzed (Participants) | 46 | 51 | 26 | 22
  Week 52 | -0.8 [-3.5 to 2.0] | 0.7 [-3.0 to 4.4] | 8.7 [-7.5 to 25.0] | 0.9 [-6.7 to 8.6]

11. Secondary Outcome: Change From Baseline in Fasting Insulin at Week 4, 12, 24 and 52
Description: Fasting Insulin, a soluble biomarker of Dysglycemia was determined in fasting blood samples to evaluate the effect of secukinumab on Dysglycemia.
Time Frame: Baseline, Week 4, 12, 24 and 52
Population: The analysis was performed in FAS population. Here, "Number analyzed" signifies participants evaluable for Fasting Insulin of Dysglycemia at week 4, 12, 24 and 52 for each arm, respectively.
Measure: Mean (95% Confidence Interval); unit: micro units per millilitre (uU/mL)
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Number analyzed (Participants) | 48 | 54 | 26 | 23
micro units per millilitre (uU/mL)
  Week 4: number analyzed (Participants) | 48 | 53 | 26 | 22
  Week 4 | 0.4 [-2.0 to 2.7] | 0.4 [-2.3 to 3.0] | -4.7 [-17.4 to 8.1] | -0.5 [-4.8 to 3.7]
  Week 12: number analyzed (Participants) | 48 | 52 | 26 | 22
  Week 12 | -1.4 [-5.1 to 2.4] | 1.1 [-2.7 to 4.8] | -2.2 [-9.2 to 4.7] | -0.1 [-4.9 to 4.7]
  Week 24: number analyzed (Participants) | 48 | 51 | 25 | 22
  Week 24 | -1.0 [-4.1 to 2.0] | 0.5 [-3.7 to 4.8] | -5.3 [-18.5 to 8.0] | -2.0 [-6.1 to 2.0]
  Week 52: number analyzed (Participants) | 48 | 51 | 26 | 22
  Week 52 | -0.4 [-4.3 to 3.6] | 1.5 [-1.3 to 4.2] | -1.2 [-7.5 to 5.1] | 3.0 [-5.2 to 11.3]

12. Secondary Outcome: Change From Baseline in Homeostatic Model Assessment (HOMA) Beta-cell Function at Week 4, 12, 24 and 52
Description: Homeostatic Model Assessment (HOMA) beta-cell function, a soluble biomarker of Dysglycemia was determined in fasting blood samples to evaluate the effect of secukinumab on Dysglycemia.
Time Frame: Baseline, Week 4, 12, 24 and 52
Population: The analysis was performed in FAS population. Here, "Number analyzed" signifies participants evaluable for HOMA beta-cell function of Dysglycemia at week 4, 12, 24 and 52 for each arm, respectively.
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Number analyzed (Participants) | 48 | 54 | 26 | 23
Percentage
  Week 4: number analyzed (Participants) | 42 | 51 | 24 | 21
  Week 4 | -18 [-64.7 to 28.2] | -0.2 [-25.7 to 25.3] | -28 [-88.4 to 33.0] | -8.9 [-38.5 to 20.7]
  Week 12: number analyzed (Participants) | 44 | 50 | 23 | 22
  Week 12 | -16 [-74.4 to 41.5] | 3.9 [-32.0 to 39.8] | -29 [-100 to 41.6] | 16.6 [-20.6 to 53.8]
  Week 24: number analyzed (Participants) | 44 | 50 | 24 | 22
  Week 24 | -25 [-53.9 to 3.5] | -8.2 [-40.2 to 23.9] | -35 [-111 to 40.7] | -26 [-63.2 to 12.0]
  Week 52: number analyzed (Participants) | 43 | 50 | 25 | 22
  Week 52 | 11.5 [-40.5 to 63.5] | -1.6 [-32.6 to 29.4] | 9.3 [-56.4 to 75.1] | 11.6 [-26.6 to 49.7]

13. Secondary Outcome: Change From Baseline in Homeostatic Model Assessment (HOMA) Insulin Resistance at Week 4, 12, 24 and 52
Description: HOMA insulin resistance, a soluble biomarker of Dysglycemia was determined in fasting blood samples to evaluate the effect of secukinumab on Dysglycemia.
Time Frame: Baseline, Week 4, 12, 24 and 52
Population: The analysis was performed in FAS population. Here, "Number analyzed" signifies participants evaluable for HOMA insulin resistance of Dysglycemia at week 4, 12, 24 and 52 for each arm, respectively.
Measure: Mean (95% Confidence Interval); unit: Insulin Resistance Index
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Number analyzed (Participants) | 48 | 54 | 26 | 23
Insulin Resistance Index
  Week 4: number analyzed (Participants) | 42 | 51 | 24 | 21
  Week 4 | 0.3 [-0.6 to 1.2] | 0.1 [-0.9 to 1.0] | -1.1 [-5.2 to 3.1] | -0.3 [-2.0 to 1.3]
  Week 12: number analyzed (Participants) | 44 | 50 | 23 | 22
  Week 12 | -0.1 [-1.5 to 1.4] | 0.6 [-0.7 to 1.8] | -0.1 [-2.5 to 2.3] | -0.4 [-2.0 to 1.3]
  Week 24: number analyzed (Participants) | 44 | 50 | 24 | 22
  Week 24 | -0.3 [-1.1 to 0.6] | 0.6 [-1.3 to 2.5] | -1.1 [-5.0 to 2.8] | -0.7 [-2.2 to 0.8]
  Week 52: number analyzed (Participants) | 43 | 50 | 25 | 22
  Week 52 | -0.2 [-1.2 to 0.9] | 0.6 [-0.3 to 1.4] | -0.2 [-2.8 to 2.4] | 0.7 [-1.9 to 3.4]

14. Secondary Outcome: Change From Baseline in Hemoglobin A1c (Glycated Hemoglobin) at Week 4, 12, 24 and 52
Description: Hemoglobin A1c (glycated hemoglobin), a soluble biomarker of Dysglycemia was determined in fasting blood samples to evaluate the effect of secukinumab on Dysglycemia.
Time Frame: Baseline, Week 4, 12, 24 and 52
Population: The analysis was performed in FAS population. Here, "Number analyzed" signifies participants evaluable for Hemoglobin A1c of Dysglycemia at week 4, 12, 24 and 52 for each arm, respectively.
Measure: Mean (95% Confidence Interval); unit: millimole per mole of Haemoglobin
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Number analyzed (Participants) | 48 | 54 | 26 | 23
millimole per mole of Haemoglobin
  Week 4: number analyzed (Participants) | 48 | 52 | 26 | 22
  Week 4 | 0.2 [-0.5 to 0.8] | -0.4 [-1.0 to 0.3] | -0.7 [-2.3 to 1.0] | -0.4 [-1.2 to 0.4]
  Week 12: number analyzed (Participants) | 48 | 54 | 26 | 22
  Week 12 | 0.4 [-0.7 to 1.5] | -0.4 [-2.2 to 1.4] | -1.2 [-3.8 to 1.3] | 0.1 [-0.8 to 1.0]
  Week 24: number analyzed (Participants) | 48 | 52 | 25 | 22
  Week 24 | -0.4 [-1.7 to 1.0] | -1.2 [-2.9 to 0.5] | -0.1 [-2.4 to 2.1] | -1.2 [-2.9 to 0.6]
  Week 52: number analyzed (Participants) | 48 | 52 | 26 | 22
  Week 52 | -1.1 [-2.3 to 0.1] | -2.8 [-6.1 to 0.4] | -1.9 [-4.3 to 0.6] | -2.1 [-3.0 to 1.2]

15. Secondary Outcome: Change From Baseline in Sex Hormone-binding Globulin (SHBG) at Week 4, 12, 24 and 52
Description: Sex hormone-binding globulin (SHBG), a soluble biomarker of Dysglycemia was determined in fasting blood samples to evaluate the effect of secukinumab on Dysglycemia.
Time Frame: Baseline, Week 4, 12, 24 and 52
Population: The analysis was performed in FAS population. Here, "Number analyzed" signifies participants evaluable for SHBG of Dysglycemia at week 4, 12, 24 and 52 for each arm, respectively.
Measure: Mean (95% Confidence Interval); unit: nanomole per Liter (nmol/L)
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Number analyzed (Participants) | 48 | 54 | 26 | 23
nanomole per Liter (nmol/L)
  Week 4: number analyzed (Participants) | 48 | 53 | 26 | 21
  Week 4 | 0.1 [-1.8 to 2.1] | 3.7 [-3.0 to 10.4] | 4.7 [-4.2 to 13.5] | -0.3 [-4.0 to 3.5]
  Week 12: number analyzed (Participants) | 48 | 54 | 26 | 21
  Week 12 | -0.1 [-3.4 to 3.2] | 1.1 [-1.8 to 4.1] | 3.7 [-1.6 to 9.1] | 4.1 [-0.2 to 8.4]
  Week 24: number analyzed (Participants) | 48 | 52 | 25 | 21
  Week 24 | -1.5 [-5.1 to 2.2] | 3.2 [-0.9 to 7.2] | 1.7 [-2.9 to 6.3] | 2.6 [-1.5 to 6.7]
  Week 52: number analyzed (Participants) | 48 | 50 | 26 | 20
  Week 52 | -3.1 [-10.8 to 4.6] | 5.9 [-1.3 to 13.0] | -2.6 [-14.9 to 9.6] | 3.2 [-4.3 to 10.8]

16. Secondary Outcome: Change From Baseline in Triglycerides, Total Cholesterol, Low Density Lipoprotein (LDL), High Density Lipoprotein (HDL), Apolipoprotein A-1 (ApoA-1) and Apolipoprotein B (ApoB) at Week 4, 12, 24 and 52
Description: Triglycerides, Total cholesterol, Low density lipoprotein (LDL), High density lipoprotein (HDL), Apolipoprotein A-1 (ApoA-1) and Apolipoprotein B (ApoB), soluble biomarkers of impaired lipid metabolism were determined in fasting blood samples to evaluate the effect of secukinumab on impaired lipid metabolism.
Time Frame: Baseline, Week 4, 12, 24 and 52
Population: The analysis was performed in FAS population. Here, "Number analyzed" signifies participants evaluable for Triglycerides, Total cholesterol, LDL, HDL, ApoA-1 and ApoB of impaired lipid metabolism at week 4, 12, 24 and 52 for each arm, respectively.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Number analyzed (Participants) | 48 | 54 | 26 | 23
mg/dL
  Triglycerides Week 4: number analyzed (Participants) | 48 | 53 | 26 | 21
  Triglycerides Week 4 | -1.8 [-15.5 to 12.0] | 6.5 [-5.9 to 18.9] | 12.7 [-12.2 to 37.7] | 27.5 [-6.6 to 61.6]
  Triglycerides Week 12: number analyzed (Participants) | 48 | 54 | 26 | 21
  Triglycerides Week 12 | -9.3 [-20.8 to 2.3] | 4.0 [-9.3 to 17.3] | 5.9 [-32.4 to 44.2] | 2.7 [-18.3 to 23.8]
  Triglycerides Week 24: number analyzed (Participants) | 48 | 52 | 25 | 21
  Triglycerides Week 24 | 4.6 [-16.6 to 25.8] | 3.9 [-9.1 to 16.9] | 32.8 [-19.7 to 85.2] | 17.1 [-2.3 to 36.5]
  Triglycerides Week 52: number analyzed (Participants) | 48 | 50 | 26 | 20
  Triglycerides Week 52 | 64.6 [-44.0 to 173.2] | 2.6 [-11.7 to 16.9] | -6.0 [-54.3 to 42.3] | 11.9 [-8.6 to 32.3]
  Total cholesterol Week 4: number analyzed (Participants) | 48 | 53 | 26 | 21
  Total cholesterol Week 4 | 0.4 [-6.4 to 7.1] | 7.1 [1.1 to 13.2] | 4.8 [-3.2 to 12.8] | -2.7 [-10.0 to 4.7]
  Total cholesterol Week 12: number analyzed (Participants) | 48 | 54 | 26 | 21
  Total cholesterol Week 12 | 3.1 [-3.1 to 9.4] | 3.6 [-4.1 to 11.2] | 10.0 [2.8 to 17.1] | -4.2 [-11.2 to 2.8]
  Total cholesterol Week 24: number analyzed (Participants) | 48 | 52 | 25 | 21
  Total cholesterol Week 24 | 0.9 [-5.2 to 7.1] | 0.6 [-4.9 to 6.1] | 7.2 [-1.5 to 16.0] | -3.2 [-12.0 to 5.5]
  Total cholesterol Week 52: number analyzed (Participants) | 48 | 50 | 26 | 20
  Total cholesterol Week 52 | 7.8 [0.0 to 15.6] | 2.3 [-5.2 to 9.9] | 8.9 [2.1 to 15.7] | 2.9 [-5.9 to 11.7]
  LDL Week 4: number analyzed (Participants) | 48 | 53 | 26 | 21
  LDL Week 4 | 1.1 [-4.6 to 6.8] | 6.8 [0.8 to 12.8] | 5.2 [-2.0 to 12.4] | -5.6 [-12.1 to 0.8]
  LDL Week 12: number analyzed (Participants) | 48 | 54 | 26 | 21
  LDL Week 12 | 2.9 [-2.2 to 7.9] | 2.7 [-4.8 to 10.1] | 9.5 [3.4 to 15.5] | -5.6 [-12.7 to 1.5]
  LDL Week 24: number analyzed (Participants) | 48 | 52 | 25 | 21
  LDL Week 24 | -2.7 [-8.1 to 2.7] | -1.3 [-6.9 to 4.4] | 1.1 [-7.4 to 9.5] | -11 [-18.9 to -2.4]
  LDL Week 52: number analyzed (Participants) | 48 | 50 | 26 | 20
  LDL Week 52 | 1.7 [-6.5 to 9.9] | -0.9 [-8.4 to 6.5] | 8.2 [1.3 to 15.0] | 1.1 [-8.4 to 10.5]
  HDL Week 4: number analyzed (Participants) | 48 | 53 | 26 | 21
  HDL Week 4 | -0.6 [-2.6 to 1.3] | 0.4 [-1.5 to 2.2] | 0.3 [-2.3 to 2.9] | -1.3 [-4.6 to 2.0]
  HDL Week 12: number analyzed (Participants) | 48 | 54 | 26 | 21
  HDL Week 12 | -0.4 [-2.4 to 1.6] | 0.2 [-1.8 to 2.2] | 1.0 [-1.2 to 3.3] | -0.5 [-4.9 to 3.8]
  HDL Week 24: number analyzed (Participants) | 48 | 52 | 25 | 21
  HDL Week 24 | 1.2 [-1.5 to 3.9] | 0.3 [-2.3 to 2.8] | -1.1 [-3.4 to 1.3] | 0.5 [-4.1 to 5.1]
  HDL Week 52: number analyzed (Participants) | 48 | 50 | 26 | 20
  HDL Week 52 | 0.1 [-2.1 to 2.4] | 1.8 [-0.5 to 4.2] | -0.3 [-2.9 to 2.4] | -1.4 [-4.6 to 1.8]
  ApoA-1 Week 4: number analyzed (Participants) | 48 | 53 | 26 | 21
  ApoA-1 Week 4 | 0.3 [-5.1 to 5.7] | 0.9 [-4.0 to 5.7] | 7.7 [-0.6 to 15.9] | -5.5 [-12.0 to 1.0]
  ApoA-1 Week 12: number analyzed (Participants) | 48 | 54 | 26 | 21
  ApoA-1 Week 12 | 4.0 [-2.0 to 10.1] | 2.4 [-1.9 to 6.8] | 7.1 [1.2 to 12.9] | -3.3 [-12.1 to 5.5]
  ApoA-1 Week 24: number analyzed (Participants) | 48 | 52 | 25 | 21
  ApoA-1 Week 24 | 5.5 [-0.9 to 12.0] | 2.8 [-3.0 to 8.6] | 3.0 [-3.3 to 9.3] | -3.1 [-11.3 to 5.1]
  ApoA-1 Week 52: number analyzed (Participants) | 48 | 50 | 26 | 20
  ApoA-1 Week 52 | -4.5 [-10.0 to 0.9] | -6.0 [-11.6 to -0.3] | -5.5 [-14.9 to 3.9] | -13 [-22.3 to -3.1]
  ApoB Week 4: number analyzed (Participants) | 48 | 53 | 26 | 21
  ApoB Week 4 | 1.5 [-2.7 to 5.6] | 3.6 [0.5 to 6.6] | 2.7 [-1.1 to 6.5] | -2.5 [-7.7 to 2.8]
  ApoB Week 12: number analyzed (Participants) | 48 | 54 | 26 | 21
  ApoB Week 12 | 4.0 [0.6 to 7.4] | 3.4 [-0.5 to 7.3] | 7.4 [3.9 to 11.0] | -1.0 [-7.0 to 4.9]
  ApoB Week 24: number analyzed (Participants) | 48 | 52 | 25 | 21
  ApoB Week 24 | 1.0 [-2.8 to 4.8] | 2.0 [-1.3 to 5.3] | 5.6 [1.4 to 9.9] | -4.2 [-10.7 to 2.3]
  ApoB Week 52: number analyzed (Participants) | 48 | 50 | 26 | 20
  ApoB Week 52 | 3.7 [-2.2 to 9.6] | 2.3 [-1.8 to 6.4] | 6.7 [3.0 to 10.5] | -0.2 [-5.4 to 5.0]

17. Secondary Outcome: Change From Baseline in Adiponectin at Week 4, 12, 24 and 52
Description: Adiponectin, a soluble biomarker of impaired lipid metabolism was determined in fasting blood samples to evaluate the effect of secukinumab on systemic inflammation.
Time Frame: Baseline, Week 4, 12, 24 and 52
Population: The analysis was performed in FAS population. Here, "Number analyzed" signifies participants evaluable for Adiponectin of impaired lipid metabolism at week 4, 12, 24 and 52 for each arm, respectively.
Measure: Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Number analyzed (Participants) | 48 | 54 | 26 | 23
ug/mL
  Week 4: number analyzed (Participants) | 48 | 53 | 26 | 22
  Week 4 | -0.5 [-1.0 to -0.1] | 0.2 [-0.4 to 0.8] | -0.1 [-0.8 to 0.5] | -0.6 [-1.2 to -0.0]
  Week 12: number analyzed (Participants) | 48 | 52 | 26 | 22
  Week 12 | -0.5 [-1.1 to -0.0] | -0.2 [-0.7 to 0.3] | 0.5 [0.1 to 0.9] | 0.3 [-0.7 to 1.3]
  Week 24: number analyzed (Participants) | 48 | 51 | 25 | 22
  Week 24 | 0.3 [-0.3 to 0.9] | 0.1 [-0.5 to 0.7] | 0.7 [-0.3 to 1.8] | -0.6 [-1.6 to 0.3]
  Week 52: number analyzed (Participants) | 48 | 51 | 26 | 22
  Week 52 | -1.1 [-1.6 to -0.6] | -0.9 [-1.5 to -0.3] | -0.4 [-1.0 to 0.2] | -1.1 [-2.0 to -0.3]

18. Secondary Outcome: Change From Baseline in Leptin at Week 4, 12, 24 and 52
Description: Leptin, a soluble biomarker of impaired lipid metabolism was determined in fasting blood samples to evaluate the effect of secukinumab on systemic inflammation.
Time Frame: Baseline, Week 4, 12, 24 and 52
Population: The analysis was performed in FAS population. Here, "Number analyzed" signifies participants evaluable for Leptin of impaired lipid metabolism at week 4, 12, 24 and 52 for each arm, respectively
Measure: Mean (95% Confidence Interval); unit: ng/mL (nanogram per milliliter)
Arm/Group | Secukinumab 300 mg | Secukinumab 150 mg | Placebo Followed by 300 mg Secukinumab | Placebo Followed by 150 mg Secukinumab
Number analyzed (Participants) | 48 | 54 | 26 | 23
ng/mL (nanogram per milliliter)
  Week 4: number analyzed (Participants) | 48 | 53 | 26 | 22
  Week 4 | -0.6 [-1.8 to 0.7] | 1.0 [-0.1 to 2.2] | -0.2 [-1.6 to 1.2] | 0.3 [-1.2 to 1.9]
  Week 12: number analyzed (Participants) | 48 | 52 | 26 | 22
  Week 12 | 0.2 [-0.7 to 1.1] | 0.1 [-0.9 to 1.2] | 0.7 [-1.0 to 2.4] | -0.3 [-1.7 to 1.2]
  Week 24: number analyzed (Participants) | 48 | 51 | 25 | 22
  Week 24 | 0.2 [-0.7 to 1.2] | 1.0 [-0.5 to 2.4] | -0.3 [-2.8 to 2.3] | -1.4 [-4.9 to 2.1]
  Week 52: number analyzed (Participants) | 48 | 51 | 26 | 22
  Week 52 | 0.2 [-1.0 to 1.3] | -0.5 [-1.6 to 0.7] | -0.4 [-3.8 to 3.0] | -2.9 [-5.7 to 0.0]

ADVERSE EVENTS:
Time Frame: From signing of Informed Consent up to 30 days post last drug treatment.
Groups:
- Secukinumab (300 mg) up to Week 12: Participants were administered with 300 mg secukinumab s.c. using pre-filled syringe every week for 4 weeks followed by 300 mg secukinumab up to 12 weeks.
- Secukinumab (150 mg) up to Week 12: Participants were administered with 150 mg secukinumab s.c. using pre-filled syringe every week for 4 weeks followed by 150 mg secukinumab up to 12 weeks.
- Placebo up to Week 12: Participants were administered with placebo up to 12 weeks.
- Secukinumab (300 mg) After Week 12: Participants were administered with 300 mg secukinumab s.c. using pre-filled syringe every week for 4 weeks followed by 300 mg secukinumab every 4 weeks until week 48 (last injection).
- Secukinumab (150 mg) After Week 12: Participants were administered with 150 mg secukinumab s.c. using pre-filled syringe every week for 4 weeks followed by 150 mg secukinumab every 4 weeks until week 48 (last injection).
- Placebo Followed by Secukinumab (300 mg) After Week 12: Participants were administered with placebo until week 12 followed by 300 mg secukinumab s.c. using prefilled syringe every week for 4 weeks followed by 300 mg secukinumab every 4 weeks until week 48 (last injection).
- Placebo Followed by Secukinumab (150 mg) After Week 12: Participants were administered with placebo until week 12 followed by 150 mg secukinumab s.c. using prefilled syringe every week for 4 weeks followed by 150 mg secukinumab every 4 weeks until week 48 (last injection).
Arm/Group | Secukinumab (300 mg) up to Week 12 | Secukinumab (150 mg) up to Week 12 | Placebo up to Week 12 | Secukinumab (300 mg) After Week 12 | Secukinumab (150 mg) After Week 12 | Placebo Followed by Secukinumab (300 mg) After Week 12 | Placebo Followed by Secukinumab (150 mg) After Week 12
Serious Adverse Events (participants affected / at risk) | 1/48 | 0/54 | 2/49 | 6/48 | 6/54 | 0/26 | 1/23
Other Adverse Events (participants affected / at risk) | 29/48 | 36/54 | 35/49 | 36/48 | 43/54 | 21/26 | 19/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (300 mg) up to Week 12 (N=48) | Secukinumab (150 mg) up to Week 12 (N=54) | Placebo up to Week 12 (N=49) | Secukinumab (300 mg) After Week 12 (N=48) | Secukinumab (150 mg) After Week 12 (N=54) | Placebo Followed by Secukinumab (300 mg) After Week 12 (N=26) | Placebo Followed by Secukinumab (150 mg) After Week 12 (N=23)
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
COLITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
DUODENAL ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
ANAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
ERYSIPELAS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
HELICOBACTER INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
PNEUMONIA BACTERIAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
VERTEBRAL FORAMINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
UTERINE POLYP (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab (300 mg) up to Week 12 (N=48) | Secukinumab (150 mg) up to Week 12 (N=54) | Placebo up to Week 12 (N=49) | Secukinumab (300 mg) After Week 12 (N=48) | Secukinumab (150 mg) After Week 12 (N=54) | Placebo Followed by Secukinumab (300 mg) After Week 12 (N=26) | Placebo Followed by Secukinumab (150 mg) After Week 12 (N=23)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
CONJUNCTIVITIS ALLERGIC (Eye disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
DRY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
EYE SWELLING (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
BURNING MOUTH SYNDROME (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 3 | 3 | 1
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
GLOSSITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1 | 1 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 0
FATIGUE (General disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0
INJECTION SITE PAIN (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
BRONCHITIS (Infections and infestations) | 1 | 1 | 0 | 3 | 1 | 0 | 0
CANDIDA INFECTION (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
CONJUNCTIVITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0
ECTHYMA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
FUNGAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 2 | 0 | 0 | 0 | 2 | 0 | 0
GASTROINTESTINAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 2 | 2 | 0 | 0
GINGIVITIS (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 1
HORDEOLUM (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 0
IMPETIGO (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
LARYNGITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 10 | 14 | 18 | 21 | 25 | 10 | 10
ORAL CANDIDIASIS (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 0
ORAL HERPES (Infections and infestations) | 0 | 2 | 0 | 2 | 2 | 1 | 1
OTITIS EXTERNA (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 0
OTITIS MEDIA (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
PARONYCHIA (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
PERIODONTITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 3 | 1 | 0
PHARYNGITIS (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
PULPITIS DENTAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
RHINITIS (Infections and infestations) | 1 | 0 | 2 | 2 | 3 | 1 | 4
ROOT CANAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
SINUSITIS (Infections and infestations) | 2 | 1 | 0 | 0 | 2 | 0 | 0
SKIN CANDIDA (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 2 | 1 | 1 | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 3 | 1 | 1 | 1 | 0 | 1
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 1 | 1
BURNS FIRST DEGREE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
BURSA INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1 | 0 | 0 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3 | 0 | 1 | 1
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 2 | 5 | 5 | 3 | 0 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 4 | 4 | 5 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 2 | 1 | 1
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
PYOGENIC GRANULOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1 | 0 | 1 | 1
DIZZINESS (Nervous system disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 0
HEADACHE (Nervous system disorders) | 4 | 6 | 2 | 7 | 7 | 2 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 2 | 2 | 0 | 1 | 0 | 2 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
MENOPAUSAL SYMPTOMS (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 2 | 4 | 1 | 0
NASAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 3 | 1 | 0
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 1 | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
INTERTRIGO (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
PAPULE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 2 | 2 | 1 | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2 | 1 | 0 | 1
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
SKIN REACTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 1 | 1 | 1 | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.